CLINICAL TRIAL: NCT04211233
Title: Diagnostic Subdural EEG-electrode And Subdural hEmatoma (DISEASE): Study Protocol for Prospective Non-randomized Controlled Trial
Brief Title: Diagnostic Subdural EEG-electrode And Subdural hEmatoma (DISEASE)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinic Frankfurt (Other)
Responsible Party: Principal Investigator, Juergen Konczalla, Pincipal Investigator, University Clinic Frankfurt
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DISEASE
Record Dates: First submitted 2019-12-18; First posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Seizures; Subdural Hematoma
Keywords: invasive grid electrode; functional outcome; predictors for seizures
MeSH Terms: conditions — Seizures; Hematoma, Subdural

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Invasive subdural arm (Active Comparator): Implantation of invasive subdural electrode in patients after surgical treatment of acute subdural hematoma
  Interventions: Device: invasive subdural grid electrode
- Standard treatment arm (Sham Comparator): Patients with acute subdural hematoma who underwent surgical Treatment and receive Standard medical treatment
  Interventions: Other: Control arm

INTERVENTIONS:
Device: invasive subdural grid electrode — A subdural EEG-electrode (PLATIN 1x4 or 1x6; Ad-Tech Medical Instrument Corporation, Oak Creek, WI, USA, Figure 1) will be implanted in the subdural space frontotemporal intraoperatively and diverted separately from the wound area. Afterwards, invasive Monitoring will be performed for 7 days and the grid will be removed simply by pulling out.
  Arms: Invasive subdural arm
Other: Control arm — Standard Treatment based on Brain Trauma Foundation
  Arms: Standard treatment arm

SUMMARY:
Epileptic seizures are one of the frequent complications in patients with traumatic brain injury; the incidence lies approximately at 20%. Particularly, acute subdural hematoma (aSDH) is one of the most important predictors for epileptic seizures, which is besides other parameters like age, preoperative Glasgow coma scale, cerebral herniation, hematoma volume and time to operation, associated with worse neurological outcome. In a recent systematic review, the mean incidence of epileptic seizures in aSDH was 28%, whereas one retrospective study focusing on EEG-diagnostic reported very high incidence of epileptiform abnormalities on surface EEG in 87% of patients with aSDH, wherefore the question rises, if the incidence of epileptic seizures is underestimated.

Despite successful evacuation of subdural hematoma, approximately one third of patients show no clinical improvement without medical explanation. Routinely, surface spot EEG is performed to detect epileptic seizures; however the sensitivity is limited due to the skin-bone barrier and the short duration of recording. Furthermore, surface EEG is not always available, for example during the night or at weekends, which is an additional limitation for the loss of treatment timing as well. Spot surface EEG will record for only 20 to 30 minutes in contrast to continuous EEG recordings that are performed for hours or days.

Due to the clinical relevance of epileptic seizures, several studies investigated the benefit of prophylactic antiepileptic treatment. To date, there is only one recommendation from the Brain Trauma Foundation at evidence class II to treat patients with severe traumatic brain injury with prophylactic antiepileptic treatment during the first week. Beyond the interval; there was no clinical benefit for patients selected. Still, there are some limitations´wherefore the clinical use of prophylactic antiepileptic treatment varies between clinicians and countries. At that time, the standard medication was phenytoin which has several side effects, but to date, there are several new intravenous antiepileptic drugs with comparable effect but better safety profile. On the other hand, there was no sifferentiation made between high-risked seizure prone patients, like patients with aSDH, and low-risked patients which is one of the limiting factors to support a general recommendation. Therefore the role of prophylactic antiepileptic treatment is still questionable.

In the clinical routine, invasive EEG-electrodes are commonly used to detect epileptic focus. The benefit of those electrodes is the real time analysis in case of seizure occurrence compared to surface EEG. Moreover, therapeutic effect is directly visible through the monitoring. Therefore the idea of this study was to make a real time analysis possible for patient with TBI, particularly aSDH, to have diagnostic and therapeutic real time monitoring detecting subclinical seizures.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged ≥18 years)
* Symptomatic aSDH needing operative treatment via craniotomy or craniectomy
* Informed consent

Exclusion Criteria:

* Patients with infaust prognosis
* Asymptomatic patients with conservative treatment
* aSDH as a secondary diagnosis
* Concurrent enrollment in any other trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-12-20 (Estimated); Primary Completion 2020-12-20 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Time-to-Seizure | up to 14 days
  The time until seizure occurrence will be compared between both arms.
Incidence of seizure | 1-7 days
  Incidence of seizures will be compared between both arms.

SECONDARY OUTCOMES:
Modified rankin scale at discharge and follow-up | 3-6 months
  Modified Rankin Scale:
  0 - No symptoms.
  1. - No significant disability.
  2. - Slight disability.
  3. - Moderate disability.
  4. - Moderately severe disability.
  5. - Severe disability.
  6. - Dead.
Glasgow outcome scale at discharge and follow-up | 3-6months
  Glasgow Outcome scale:
  1. Death
  2. Persistent vegetative state
  3. Severe disability
  4. Moderate disability
  5. Low disability

CONTACTS AND LOCATIONS:
Locations (1):
- Goethe University Hospital, Frankfurt am Main, Germany

IPD SHARING:
Plan to Share IPD: Undecided
email contact.

REFERENCES:
- [Derived] Won SY, Freiman TM, Reif PS, Dubinski D, Hattingen E, Herrmann E, Seifert V, Rosenow F, Strzelczyk A, Konczalla J. DIagnostic Subdural EEG electrodes And Subdural hEmatoma (DISEASE): a study protocol for a prospective nonrandomized controlled trial. Neurol Res Pract. 2020 Dec 15;2:50. doi: 10.1186/s42466-020-00096-8. eCollection 2020. PMID 33344885